CLINICAL TRIAL: NCT03885674
Title: Improving Medication Self-Administration and Health After Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, A. M. Barrett, MD, Director, Center for Stroke Rehabilitation Research, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-623-08; CBIR161RG041 (Other Grant/Funding Number: New Jersey Commission on Brain Injury Research)
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Stroke; Stroke, Acute; Cognitive Impairment; Brain Injuries, Traumatic; Medication Adherence; Medication Compliance
MeSH Terms: conditions — Stroke; Cognitive Dysfunction; Brain Injuries, Traumatic; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of three intervention groups; video call reminders, automated text messages, or no intervention (standard care).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reminder Interventions (Experimental): Receive daily reminders from Kessler Foundation study personnel on when to take their medication.
  Interventions: Other: Video Call Reminder Condition; Other: Automated Text Message Reminder Condition
- Standard Condition (No Intervention): This group will not receive reminders on when to take their medication from Kessler Foundation staff and will receive the usual and standard care.

INTERVENTIONS:
Other: Video Call Reminder Condition — Receive daily video call reminders from Kessler Foundation research staff directly at the time of each medication dose and instructed to take the medication while on the video call.
  Arms: Reminder Interventions
Other: Automated Text Message Reminder Condition — Receive daily automated text messages at the time of each medication dose and will be instructed to take the medication at that time. Each text message reminder will also contain a photo of the medication to be taken. On a weekly basis, study personnel will contact participants in this group to make sure they are receiving the text messages appropriately.
  Arms: Reminder Interventions

SUMMARY:
The purpose of this research study is to assess medication self-administration (MSA) and the impact of three different interventions on improving medication adherence. The findings for this study may help develop evidence-based reminder protocols to reduce medication self-administration errors after brain injury.

DETAILED DESCRIPTION:
The investigators are interested in studying how brain injury (TBI, stroke, etc.) survivors manage self-administering their medication once they return home, and are aiming to improve their medication adherence. In this six month long study, patients will be placed into one of three intervention groups 1) standard care received (usual care, no reminder provided), 2) receive a video call at time medication is to be taken, 3) receive an automated text message when medication is to be taken. The investigators aim to identify which intervention is best at helping brain injury survivors adhere to their medication schedule, with the future goal of implementing this type of reminder protocol into standard care.

Hypothesis: The investigators hypothesize that automated reminder text messages will result in MSA improvement comparable to video calls, maintained over the six month period.

Allocation to groups: Patients will be randomized to receive video calls, automated text messages, or no intervention (standard care). The randomization schedule is by computer-generated number list.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18
* Less than three months post Brain Injury event
* English speaking (learned English at age 10 or younger, and use it daily)
* Currently taking up to eight medications on a daily basis

Exclusion Criteria:

* Legally blind
* Unable to give informed consent due to comprehension deficits
* Severe memory or cognitive impairments that would not allow for formal testing, as determined by the investigator
* History of psychiatric hospitalization for attempted overdose of pills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | 6 months
  As measured by Medication Event Monitoring System (MEMS) trackers

CONTACTS AND LOCATIONS:
Overall Officials: AM Barrett, MD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrett AM, Galletta EE, Zhang J, Masmela JR, Adler US. Stroke survivors over-estimate their medication self-administration (MSA) ability, predicting memory loss. Brain Inj. 2014;28(10):1328-33. doi: 10.3109/02699052.2014.915984. Epub 2014 Jun 2. PMID 24884398